CLINICAL TRIAL: NCT06249464
Title: A Random Controlled Study to Explore the Effect of Stellate Ganglion Block on Pharyngeal Dysphagia After Cerebralvascular Accident
Brief Title: Effect of Stellate Ganglion Block on Pharyngeal Dysphagia After Cerebralvascular Accident
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Principle Investigator, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGB for stroke old
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate Ganglion Block group (Experimental): Patients enrolled were firstly numbered for privacy with software and divided into the observation group (n=33) and the control group (n=33) with a random number table. Additionally, the staffs involved in assessment would not participate in the intervention of the study. The treatment lasted 20 days.
  Interventions: Behavioral: comprehensive rehabilitation; Drug: Lidocaine hydrochloride
- Routine treatment group (Active Comparator): Patients enrolled were firstly numbered for privacy with software and divided into the observation group (n=33) and the control group (n=33) with a random number table. Additionally, the staffs involved in assessment would not participate in the intervention of the study. The treatment lasted 20 days.
  Interventions: Behavioral: comprehensive rehabilitation

INTERVENTIONS:
Behavioral: comprehensive rehabilitation — All the participants were provided with the comprehensive rehabilitation (routine rehabilitation and swallowing function training). The routine rehabilitation included intervention for risk factors (blood pressure, blood lipids, blood glucose, smoking and alcohol restriction, exercise, etc.) and pharmacological treatment (aspirin, statins, anticoagulants, etc.).
  Regrading swallowing function training, both groups were given swallowing function training, including 1) exercises of closure of the vocal folds, pharyngeal, and laryngeal muscles exercises, and respiratory muscle strength training, for 15 min each time and twice per day. 2) isotonic／isometric swallowing exercises, supraglottic swallowing exercises, and the Mendelsohn maneuver, for 20 min each time and twice per day. 3) effortful swallowing exercises, and cough reflex training, for 10 min each time and twice per day.
Drug: Lidocaine hydrochloride — the observation group was given SGB once a day, with 10 sessions as a course of treatment and each side of the body for one course. All the materials included: 1) 1.5ml of 2% Lidocaine hydrochloride injection (1ml: 0.5mg), Vitamin B12 Injection 500ug (1ml: 0.5g), the 5 ml disposable syringe and the sterile disposable dental injection needles. The specific operation procedure was as follows[16]: The operator stood at the patient's block side, and the patient was placed in the supine position, with the head leaning 45 degrees toward the contralateral side of the block side. After routine disinfection of the skin, a paratracheal approach was adopted, which was, 2.5cm above the sternoclavicular joint and 1.5cm outside the midline of the neck.
  Arms: Stellate Ganglion Block group

SUMMARY:
This was a multicenter randomized controlled study. 66 post-stroke patients with pharyngeal dysphagia were randomly allocated to the observation group (n=33) or the control group (n=33). Both groups were provided with comprehensive rehabilitation including routine rehabilitation and swallowing function training. Besides, the observation group additionally underwent the stellate ganglion block (SGB). At admission and after 20-day treatment, Kubota water swallowing test, video fluoroscopic swallowing study (VFSS), and Rosenbek penetration-aspiration scale (PAS) were used to assess swallowing function.

DETAILED DESCRIPTION:
Dysphagia is a frequent and potentially serious complication of stroke. However, there is no effective measure for the treatment of pharyngeal dysphagia in stroke patients. This study aims to explore the efficacy of stellate ganglion block in post-stroke pharyngeal dysphagic patients who received comprehensive rehabilitation. This was a multicenter randomized controlled study. 66 post-stroke patients with pharyngeal dysphagia were randomly allocated to the observation group (n=33) or the control group (n=33). Both groups were provided with comprehensive rehabilitation including routine rehabilitation and swallowing function training. Besides, the observation group additionally underwent the stellate ganglion block (SGB). At admission and after 20-day treatment, Kubota water swallowing test, video fluoroscopic swallowing study (VFSS), and Rosenbek penetration-aspiration scale (PAS) were used to assess swallowing function.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 80 years;
* New-onset stroke;
* The course of disease between 1 to 6 months;
* With pharyngeal dysphagia;
* Stable vital signs;
* Voluntary participation in the study.

Exclusion Criteria:

* Allergy to Lidocaine injection or vitamin B12 injection;
* Severe cognitive impairment;
* Coagulation disorders;
* Severe dysfunction of organs including heart, lungs, kidney, liver, etc.;
* Complicated with other neurological diseases;
* Dysphagia caused by other diseases or reasons.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Video fluoroscopic swallowing study | day 1 and day 20
  The patient was required to take a sitting position with the head naturally upright. Under the guidance of the examiner, the patient first swallowed 5ml of iohexol solution (50ml:17.5g in iodine terms). If the patient exhibited aspiration, the test would stop. If not, the patient was instructed to swallow 10ml of iohexol solution mixed with breadcrumbs, and the patient's swallowing condition was observed with immediate measures ready to take for safety. Specially, the esophageal phase was not included in the study, because it was commonly regarded as an independent phase. The swallowing were divided into 3 phases in this assessment: Oral phase, Pharyngeal phase, and Aspiration, with maximum 3,3,4 points were given to each phase. The total score was calculated as the final result. The final score was positively correlated with the swallowing function.

SECONDARY OUTCOMES:
Kubota water swallowing test | day 1 and day 20
  During the test, patients were required to drink 30 ml of warm water. According to the situation, the swallowing function was rated from Level 1 (excellent) to Level 5 (poor). Specifically, Grade 1: The patient drank all the water at once without choking; Grade II: The patient drank all the water in two or more times without choking; Grade III: The patient drank all the water at once with choking; Grade IV: The patient drank all the water in two or more times with choking; Grade V: The patient exhibited difficulty drinking with frequent choking.
penetration-aspiration scale | day 1 and day 20
  this assessment evaluated the patient's swallowing of contrast medium and whether there was retention, penetration, and aspiration. It included multiple items, each with the corresponding criteria, Specifically, whether the swallowed material entered the airway, passed through or contacted the vocal cords, and whether the patient exhibited the corresponding ability to clear. There were 8 levels in the results, with higher levels indicating more severe aspiration.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Xinzhu Rehabilitation Hospital, Xinzhu, Taiwan

IPD SHARING:
Plan to Share IPD: No